CLINICAL TRIAL: NCT04820426
Title: Evaluation of the Effect of Neuropathic Pain on Quality of Life in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, YILDIZ GONCA DOGRU, Resident of Physical Medicine and Rehabilitation, Ahi Evran University Education and Research Hospital
Other Study IDs: 2021-06/55
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis; Neuropathic Pain
Keywords: rheumatoid arthritis; neuropathic pain; pain in rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis patients: Rheumatoid arthritis patients will be evaluated in terms of the presence of neuropathic pain and its effect on the quality of life, at their admission.

SUMMARY:
Rheumatoid arthritis is a chronic inflammatory disease that mainly affects the joint synovium. Rheumatoid arthritis patients define pain as their major symptom and the most important reason for applying to a healthcare institution. Approximately 70% of rheumatoid arthritis patients state that improvement in their pain compared to other symptoms of the disease is their priority. Pain in rheumatoid arthritis patients is also important as the disease affects approximately 0.5-1% of patients worldwide.

Although pain in rheumatoid arthritis patients can be persistent or intermittent, localized or widespread, it has often been associated with fatigue and psychosocial stress. Although nociceptive pain,defined as 'gnawing' or 'aching', is frequently observed in rheumatoid arthritis patients, typical neuropathic pain,such as 'burning' or 'itching', can be observed in some RA patients. It is thought that neuropathic pain may occur as a result of lesions or disease affecting the somatosensorial nervous system. Neuropathic pain can occur with little or no stimulus, and its symptoms are abnormal sensations such as hyperalgesia and allodynia.

The diagnosis and treatment of neuropathic pain in rheumatoid arthritis patients is important because neuropathic pain does not decrease with traditional disease-modifying anti-inflammatory drugs used in rheumatoid arthritis and causes a decrease in quality of life. In order to distinguish neuropathic pain from chronic pain, methods based on defining the quality of pain are often used. Some of these methods are; The McGill Pain Questionnaire, PainDETECT, RAPS (Rheumatoid Arthritis Pain Scale), VAS (visual analog scale), AIMS (Arthritis Impact Scale), EQ-5D (European Quality of Life Assessment and Pain Assessment Questionnaire).

The diagnosis and treatment of neuropathic pain in rheumatoid arthritis patients is important because neuropathic pain does not decrease with traditional disease-modifying anti-inflammatory drugs used in rheumatoid arthritis and causes a decrease in quality of life.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic inflammatory disease that mainly affects the joint synovium. Rheumatoid arthritis patients define pain as their major symptom and the most important reason for applying to a healthcare institution. Approximately 70% of rheumatoid arthritis patients state that improvement in their pain compared to other symptoms of the disease is their priority. Pain in rheumatoid arthritis patients is also important as the disease affects approximately 0.5-1% of patients worldwide.

Synovial inflammation, which can lead to joint deformity by causing cartilage and bone destruction, is the main pathophysiological mechanism in rheumatoid arthritis, and therefore the main cause of pain in rheumatoid arthritis patients is thought to be nociceptive. Although pain in rheumatoid arthritis was previously associated with tissue damage and inflammatory processes in the joints, accumulated knowledge shows that peripheral inflammation, disease progression, structural and neurochemical changes in the joints and sensorial system, and central pain process mechanisms may also play a role in these rheumatoid arthritis patients.

Although pain in rheumatoid arthritis patients can be persistent or intermittent, localized or widespread, it has often been associated with fatigue and psychosocial stress. Although nociceptive pain, defined as 'gnawing' or 'aching', is frequently observed in rheumatoid arthritis patients, typical neuropathic pain, such as 'burning' or 'itching', can be observed in some RA patients. It is thought that neuropathic pain may occur as a result of lesions or disease affecting the somatosensorial nervous system. Neuropathic pain can occur with little or no stimulus, and its symptoms are abnormal sensations such as hyperalgesia and allodynia.

Although the frequency of neuropathic pain in rheumatoid arthritis patients varies in various clinical studies, it is approximately 20.7-30%. The diagnosis and treatment of neuropathic pain in rheumatoid arthritis patients is important because neuropathic pain does not decrease with traditional disease-modifying anti-inflammatory drugs used in rheumatoid arthritis and causes a decrease in quality of life. To distinguish neuropathic pain from chronic pain, methods based on defining the quality of pain are often used. Some of these methods are; The McGill Pain Questionnaire, PainDETECT, RAPS (Rheumatoid Arthritis Pain Scale), VAS (visual analogue scale), AIMS (Arthritis Impact Scale), EQ-5D (European Quality of Life Assessment and Pain Assessment Questionnaire).

Although non-steroidal anti-inflammatory drugs(NSAIDs) are used for pain in rheumatoid arthritis, it is not suitable for long-term disease control. It is important to start the use of disease-modifying agents (DMARDs) in the early period in patients.

Analgesic agents such as NSAIDs, acetaminophen, and opioids are used for pain in rheumatoid arthritis patients. However, some side effects of these drugs frequently limit their usage. Long-term opioid use in pain treatment is not recommended due to its side effects such as constipation, nausea and vomiting, and should be used with careful monitoring when necessary. Other drugs such as tricyclic antidepressants and topical capsaicin have been used in randomized controlled trials for pain management in RA with limited success.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rheumatoid arthritis,
* who can read and write in Turkish,
* participant's admission participating in the study,
* participants who do not have exclusion criteria

Exclusion Criteria:

* participant's refusal to participate in the study,
* lack of cooperation due to cognitive impairment,
* participant's who have a neurological disease,
* presence of drug abuse,
* presence of malignancy in any organ or system,
* serious psychiatric problems (psychosis, etc.),
* the presence of another rheumatological disease other than Rheumatoid Arthritis,
* serious and unstable metabolic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of presence of neuropathic pain | Participant's admission
  With the "Mc Gill-Mellzack Pain Questionnaire" form, the location of the patients' pain, the nature and intensity of the pain and the relationship between time and pain will be questioned.
Evaluation of participant's anxiety and depression | Participant's admission
  Participant's anxiety and depression will be measured with Hospital Anxiety and Depression Scale (HADS). The Scale contains 14 questions.(7 anxiety and 7 depression) Each question is scored 0 to 3.
  8-10 scores mild, 11-14 scores moderate, 15-21 severe Anxiety and depression score will be measured separately.
Participants' quality of life assessed with Short Form-36 Scale | Participant's admission
  SF-36 scale, which is a quality of life assessment scale and has 36 questions, will be used to learn the participants' views about their own health, how they feel and how well they can perform daily activities.
Participants's body pain assessed by VAS | Participant's admission
  Pain will be questioned with Visual Analog Scale.(VAS) Visual Analog Scale is determined by measuring the distance (mm) on the 10 cm line, between anchor and the patient's mark. Providing a range of scores from 0-100.A higher score indicates greater pain intensity.
  No pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Evaluation of rheumatoid arthritis disease activity | Participant's admission
  Rheumatoid arthritis disease activity will be evaluated by DAS28-CRP (C Reactive Protein)
Evaluation of rheumatoid arthritis remission | Participant's admission
  Boolean index criteria will be used for detect the remission.

CONTACTS AND LOCATIONS:
Overall Officials: FIGEN TUNCAY, PROF.,M.D., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kirsehir Ahi Evran University Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noda K, Tajima M, Oto Y, Saitou M, Yoshiga M, Otani K, Yoshida K, Kurosaka D. How do neuropathic pain-like symptoms affect health-related quality of life among patients with rheumatoid arthritis?: A comparison of multiple pain-related parameters. Mod Rheumatol. 2020 Sep;30(5):828-834. doi: 10.1080/14397595.2019.1650462. Epub 2019 Aug 9. PMID 31398076
- [Background] Ito S, Kobayashi D, Murasawa A, Narita I, Nakazono K. An Analysis of the Neuropathic Pain Components in Rheumatoid Arthritis Patients. Intern Med. 2018 Feb 15;57(4):479-485. doi: 10.2169/internalmedicine.9235-17. Epub 2017 Dec 8. PMID 29225253
- [Background] Bas DB, Su J, Wigerblad G, Svensson CI. Pain in rheumatoid arthritis: models and mechanisms. Pain Manag. 2016;6(3):265-84. doi: 10.2217/pmt.16.4. Epub 2016 Apr 18. PMID 27086843
- [Background] Koop SM, ten Klooster PM, Vonkeman HE, Steunebrink LM, van de Laar MA. Neuropathic-like pain features and cross-sectional associations in rheumatoid arthritis. Arthritis Res Ther. 2015 Sep 3;17(1):237. doi: 10.1186/s13075-015-0761-8. PMID 26335941